CLINICAL TRIAL: NCT05978856
Title: The Accuracy of Computer Software Prediction of Soft Tissue Profile for Patients Undergoing Fixed Orthodontic Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Salah Hasan Saleh Mohamed, General Physician at the Ministry of Health, Al-Azhar University
Other Study IDs: VTO
Record Dates: First submitted 2023-07-17; First posted 2023-08-07 (Actual); Last update posted 2023-08-07 (Actual); Status verified 2023-07

CONDITIONS: Dental Malocclusion
Keywords: VTO; orthodontic software; prediction
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- A: real photoes (after treatment)
  Interventions: Other: Accuracy of computer software in predicting soft tissue profile changes
- B: simulated photoes

INTERVENTIONS:
Other: Accuracy of computer software in predicting soft tissue profile changes — Separate analyses will be performed on the initial and final cephalograms.
  * All of the cephalometric analyses will be done via computer software,the linear and angular measurements will be done via the software.
  * Through the use of software, the initial cephalogram and the initial photograph will be linked.
  * Then, the final values of some angles will be tracted from the post-treatment cephalogram.
  * These values will be inserted in the "treatment simulation"section of the software.
  * A post-treatment projected image of the patient will be simulated by the software.
  * Then the actual post-treatment photograph will be placed on the simulated image in transparent form.
  * From the pupil , real horizontal and vertical reference lines will be drawn.
  * Then certain measurements will be taken from referance lines to fixed points on the soft tissue to determine the discrepancies between the real and simulated images.
  Other Names: visual treatment objective
  Groups: A

SUMMARY:
A clinical study to evaluate the accuracy of computer software in predicting soft tissue profile changes in patients undergoing fixed orthodontic treatment

DETAILED DESCRIPTION:
The computer software programs exhibit certain soft tissue simulation . The purpose of the study to assess the accuracy of computer software in predicting profile changes in patients undergoing fixed orthodontic treatment

ELIGIBILITY:
The inclusion criteria included:

* Patient undergo fixed orthodontic treatment with the edgewise technique.
* Skeletal class I.
* Dental class I or II or III.
* Final class I occlusion without spacing or crowding, with normal overjet and overbite (2-4 mm)
* Availability of full diagnostic and therapeutic records before to and following orthodontic treatment, including medical and dental history, dental casts, panoramic and cephalometric x-rays, and photographic photographs.

The exclusion criteria included:

* Missing tooth or significant Bolton discrepancies (more than 3 mm).
* Craniofacial syndromes or skeletal abnormalities.
* Failed orthodontic treatment in the past.
* Cosmetic or reconstructive facial surgery during orthodontic treatment, or up to a year beforehand.
* Using drugs that could reduce the volume of soft tissues.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be performed on patients treate in the orthodontics department, faculty of dentistry, alazhar university,assuit branch.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
accuracy of computer software in predicting soft tissue profile changes | through study completion, an average of 1 year
  * Separate analyses will be performed on the initial and final cephalograms.
  * All of the cephalometric analyses will be done via computer software; the linear and angular measurements will be done via the software.
  * Through the use of software, the initial cephalogram and the initial photograph will be linked.
  * Then, the final values of some angles will be extracted from the post-treatment cephalogram.
  * These values will be inserted in the "treatment simulation" section of the software.
  * A post-treatment projected image of the patient will be simulated by the software.
  * Then the actual post-treatment photograph will be placed on the simulated image in transparent form.
  * From the pupil , real horizontal and vertical reference lines will be drawn.
  * Then certain measurements will be taken from reference lines to fixed points on the soft tissue to determine the discrepancies between the real and simulated images.

CONTACTS AND LOCATIONS:
Locations (1):
- Dental medicine al-azhar university, Asyut, Assuit, Egypt

REFERENCES:
- [Background] Kolokitha OE, Chatzistavrou E. Factors influencing the accuracy of cephalometric prediction of soft tissue profile changes following orthognathic surgery. J Maxillofac Oral Surg. 2012 Mar;11(1):82-90. doi: 10.1007/s12663-011-0253-6. Epub 2011 Jul 7. PMID 23450114
- [Background] Kolokitha OE. Validity of a manual soft tissue profile prediction method following mandibular setback osteotomy. Eur J Dent. 2007 Oct;1(4):202-11. PMID 19212468
- [Background] Leonardi R, Annunziata A, Licciardello V, Barbato E. Soft tissue changes following the extraction of premolars in nongrowing patients with bimaxillary protrusion. A systematic review. Angle Orthod. 2010 Jan;80(1):211-6. doi: 10.2319/010709-16.1. PMID 19852663
- [Background] Drobocky OB, Smith RJ. Changes in facial profile during orthodontic treatment with extraction of four first premolars. Am J Orthod Dentofacial Orthop. 1989 Mar;95(3):220-30. doi: 10.1016/0889-5406(89)90052-8. PMID 2923102
- [Background] Al-Omiri MK, Abu Alhaija ES. Factors affecting patient satisfaction after orthodontic treatment. Angle Orthod. 2006 May;76(3):422-31. doi: 10.1043/0003-3219(2006)076[0422:FAPSAO]2.0.CO;2. PMID 16637722
- [Background] Kolokitha OE, Topouzelis N. Cephalometric methods of prediction in orthognathic surgery. J Maxillofac Oral Surg. 2011 Sep;10(3):236-45. doi: 10.1007/s12663-011-0228-7. Epub 2011 May 17. PMID 22942594
- [Background] Smith JD, Thomas PM, Proffit WR. A comparison of current prediction imaging programs. Am J Orthod Dentofacial Orthop. 2004 May;125(5):527-36. doi: 10.1016/S0889540604001210. PMID 15127020
- [Background] Patterson Dental Supply. Imaging. In: Dolphin Imaging. 2012. Retrieved December 17th 2012, from http://www.dolphinimaging.com/imaging.html.
- [Background] Gossett CB, Preston CB, Dunford R, Lampasso J. Prediction accuracy of computer-assisted surgical visual treatment objectives as compared with conventional visual treatment objectives. J Oral Maxillofac Surg. 2005 May;63(5):609-17. doi: 10.1016/j.joms.2005.01.004. PMID 15883933
- [Background] Ioannidou-Marathiotou I, Papamanou DA, Papadopoulos MA. Orthodontics and esthetics of the face: from the "canons" of ancient times to contemporary pluralism. A critical review. Prog Orthod. 2008;9(2):20-33. PMID 19350056
- [Background] Prabhakar R, Rajakumar P, Karthikeyan MK, Saravanan R, Vikram NR, Reddy A. A hard tissue cephalometric comparative study between hand tracing and computerized tracing. J Pharm Bioallied Sci. 2014 Jul;6(Suppl 1):S101-6. doi: 10.4103/0975-7406.137401. PMID 25210347
- [Background] Nadjmi N, Tehranchi A, Azami N, Saedi B, Mollemans W. Comparison of soft-tissue profiles in Le Fort I osteotomy patients with Dolphin and Maxilim softwares. Am J Orthod Dentofacial Orthop. 2013 Nov;144(5):654-62. doi: 10.1016/j.ajodo.2013.06.019. PMID 24182581